CLINICAL TRIAL: NCT00148135
Title: A Phase II Trial Evaluating the Combination of Carboplatin, Gemcitabine, and Capecitabine in Patients With Carcinoma of Unknown Primary Site
Brief Title: Combination of Carboplatin, Gemcitabine, and Capecitabine in Patients With Carcinoma of Unknown Primary Site
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: recruitment goals met
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: UMCC 2001-021
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2008-01-10 (Estimated); Status verified 2007-12

CONDITIONS: Carcinoma of Unknown Primary
Keywords: Carcinoma of Unknown Primary Site (CUP)
MeSH Terms: conditions — Neoplasms, Unknown Primary | interventions — Carboplatin; Gemcitabine; Capecitabine

INTERVENTIONS:
Drug: Carboplatin
Drug: Gemcitabine
Drug: Capecitabine

SUMMARY:
This study is for patients with a type of cancer called carcinoma of unknown primary site (CUP), meaning that the site of the body where the tumor has originated is not clear. Currently, carcinoma of unknown primary site (CUP) accounts for about 5% of all newly diagnosed malignancies. The stage of the tumor is such that it is not treatable by surgery. Currently, the standard treatment for such a type of cancer at that stage is chemotherapy. However, the overall prognosis for patients with metastatic CUP remains poor, even if treated with conventional chemotherapy. Through ongoing research at medical centers around the world, doctors are trying to improve on the presently available chemotherapy regimens. The purpose of the investigators' study is similar: it is trying to determine whether a combination of three chemotherapy drugs - carboplatin, gemcitabine, and capecitabine - will improve the treatment of patients with metastatic CUP. The reason the investigators are interested in the above combination of chemotherapy agents is that each one of them is already used in patients with a variety of specific tumors, such as lung cancer, breast cancer, pancreatic cancer, colon cancer, etc.

This research study will help determine whether the combination of carboplatin, gemcitabine and capecitabine can be used and is effective in patients with carcinoma of unknown primary site.

DETAILED DESCRIPTION:
Carcinoma of unknown primary site (CUP) accounts for approximately 5% of all newly diagnosed malignancies. The overall prognosis for patients with CUP remains poor, with median survival less than one year with modern chemotherapy combinations and virtually no long-term survivors.

It has been recognized that patients with CUP represent a heterogeneous group of tumors. Managing patients with CUP requires a complete medical history, careful consideration of findings on physical exam, targeted radiologic studies and pathologic analysis of biopsy and/or surgical specimens. Within this heterogeneous group there exist at least four subsets of patients with CUP, that based on clinicopathologic features are treated with regimens which have demonstrated efficacy in tumors originating in the most likely primary site of that CUP; squamous carcinoma involving mid or high levels of cervical lymph nodes, women with isolated axillary adenopathy containing adenocarcinoma, women with a predominant presentation of peritoneal carcinomatosis and young men with extragonadal germ cell syndrome.

Unfortunately, a majority of patients with CUP do not fall into any of the above subsets and these represent a therapeutic dilemma, as there is no single regimen to date that has shown significant activity or has resulted in prolonged survival for these patients with particularly poor prognosis. Thus, new therapeutic combinations need to be investigated for treatment of these patients with CUP.

Platinum compounds have been the cornerstone of chemotherapy regimens for a wide variety of solid tumors, including lung, urothelial, head and neck, ovarian and endometrial carcinomas, as well as testicular carcinomas. Cisplatin and its analog carboplatin are currently used in chemotherapy combinations to treat CUP. Carboplatin has fewer non-hematologic side effects compared to cisplatin including less nausea and vomiting, peripheral neuropathy, nephrotoxicity and ototoxicity making it an attractive agent to combine with other drugs.

In recent years, new agents active in solid malignancies have been developed. Gemcitabine is one such agent. It is a deoxycytidine analogue structurally related to cytosine arabinoside. Gemcitabine is activated by deoxycytidine kinase in three steps of phosphorylation into difluorodeoxycytidine triphosphate, which when incorporated into DNA, leads to chain termination. Gemcitabine has been shown to have activity in pancreatic, breast, non-small cell lung carcinomas as well as in carcinomas of unknown primary site. Because of its mild toxicity profile, gemcitabine has been used in combination with other chemotherapy agents. There is evidence of in vitro and in vivo synergy between gemcitabine and the platinum compounds.

Capecitabine is an orally administered fluoropyrimidine that undergoes a three-step conversion into 5-FU, with pharmacokinetics that mimic low dose continuous infusion 5-FU. The oral formulation allows for convenient continuous therapy, avoiding a need for central venous catheters and external infusion pumps.

The final step of conversion of capecitabine into 5-FU is catalyzed by thymidine phosphorylase (TP), an enzyme which has been shown to be over expressed in colorectal tumors. This selective tumor activation has been demonstrated to lead to higher concentrations of 5-FU in tumor cells as compared to normal tissue, suggesting tumor targeting by the oral drug. Capecitabine was initially approved by the FDA for treatment of refractory breast carcinoma and has shown activity in metastatic colorectal carcinoma. Capecitabine is an attractive agent for use in combination chemotherapy due to its non-overlapping toxicity profile with many agents and lack of hematologic toxicity.

Gemcitabine has been combined with 5-FU, and may enhance the activity of 5-FU in vivo. Gemcitabine is an inhibitor of ribonucleotide reductase, an enzyme needed for synthesis of deoxynucleotides, and 5-FU interferes with dTTP synthesis by inhibition of thymidylate synthase (TS). It is plausible that concomitant administration of gemcitabine and capecitabine, may result in increased cytotoxicity by reducing intracellular dTTP thru two different mechanisms, thereby inhibiting DNA replication and repair. Platinum compounds lead to cell death by forming DNA adducts and causing double strand breaks. By inhibiting DNA synthesis and repair, both gemcitabine and 5-FU analogues could potentiate the activity of carboplatin. These interactions may underlie the clinical synergism that has been observed with platinum/5-FU and platinum/gemcitabine combinations.

We propose to combine carboplatin, gemcitabine and capecitabine as a palliative treatment for patients with CUP. Programs evaluating the incorporation of newer chemotherapy agents into combinations are reasonable in an attempt to improve outcome in patients with CUP. In addition to anticipated anti-tumor activity, the proposed combination provides a convenient schedule of brief intravenous treatment, the use of the oral agent capecitabine, and a toxicity profile which is expected to be mild, characteristics which are important in palliative treatment programs.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of carcinoma, with clinical evidence of metastasis and the primary site not clear after the following work-up:

  * Complete history and physical
  * Laboratory evaluation including serum beta-human chorionic gonadotropin (HCG), serum alpha-fetoprotein for undifferentiated or poorly differentiated carcinomas and serum prostate specific antigen (PSA) in men.
  * Directed radiologic evaluation including, at a minimum, computerized tomography (CT) of chest, abdomen and pelvis and bilateral mammography for female patients.
  * Pathologic immunohistochemistry studies of the surgical or biopsy specimen, including studies for estrogen receptor/progesterone receptor and PSA stains when clinically appropriate.
* Patients must be at least 18 years of age and have a Zubrod performance status 0-2.
* Adequate organ function, defined as absolute neutrophil count (ANC) > 1500/ul, platelet count of > 100,000/ul, serum creatinine less than or equal to 2.0 mg/dl, serum bilirubin less than or equal to 1.5 mg/dl.
* Patients must have measurable disease. (Partial response [PR] - at least a 30% decrease in the sum of LD of target lesions taking as reference the baseline sum LD.)
* Patients may be previously untreated or have received one chemotherapy regimen provided it did not include carboplatin, gemcitabine or capecitabine.
* Patients must have no serious intercurrent medical or psychiatric illness that would limit their ability to provide informed consent or receive protocol therapy.
* Patients must be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to the initiation of therapy.

Exclusion Criteria:

* Patients with previous invasive malignancy within the preceding 5 years are ineligible unless clinicopathologic information regarding the current neoplasm is clearly discordant from prior disease. Patients with non-melanoma skin cancer or in situ cancer of any site are eligible.
* Patients with brain metastasis are not eligible.
* No concurrent chemotherapy, biological or radiotherapy is allowed.
* Pregnant or lactating women are not eligible. Women and men of childbearing potential must agree to use effective contraception throughout the treatment period, and for six months after treatment has been discontinued.
* The following groups of patients will not be eligible for the study as they represent populations of patients with CUP for whom more specific treatment approaches are available:

  1. Patients presenting with squamous carcinoma isolated to middle and high cervical lymph nodes
  2. Women presenting with isolated axillary lymphadenopathy
  3. Women presenting with predominant peritoneal carcinomatosis
  4. Men < 50 years of age presenting with predominant mediastinal and/or retroperitoneal nodal involvement and biopsy showing undifferentiated or poorly differentiated carcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-05; Primary Completion 2006-04 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Zalupski, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States